CLINICAL TRIAL: NCT02676063
Title: Long Term Prognostic of Neonatal Hypoxic Ischemic Encephalopathy in the Era of Neuroprotective Treatment With Hypothermia
Brief Title: Long Term Prognostic of Neonatal Hypoxic Ischemic Encephalopathy With Hypothermia Treatment
Acronym: LyTONEPAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC1416
Record Dates: First submitted 2015-09-28; First posted 2016-02-08 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Ischemic-Hypoxic Encephalopathy
Keywords: predictive factors; neurodevelopmental disabilities
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neonatal Hypoxic Ischemic encephalopathy: moderate or severe HIE among term and late preterm newborn

SUMMARY:
The primary objective is to evaluate neonatal characteristics, and biological and clinical investigations as predictive factors of death, or of severe and moderate neurodevelopmental disability at 3 years, in a large population-based cohort of full-term and late preterm neonates with moderate or severe HIE.

Contrary to most previous studies which have often analyzed the accuracy of one factor among all other clinical investigations, the investigators objective's is to seek a relevant combination of several factors among the following list:

* Neonatal characteristics: gestational age and birthweight, maternal disease, acute intrapartum event, delivery mode, acidosis, neurological examination, place of birth and neonatal transfer
* Laboratory investigations: pH, lactates and new biological markers as detailed below
* Clinical investigations: aEEG, EEG, MRI, diffusion-weighted MRI

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a rare neonatal condition affecting about 1‰ births and with a high rate of death and severe neurological disability despite significant improvement of the management of this illness in the last ten years. During the first hours and days of life, different examinations are made by neonatologists to guide decisions about the management of HIE and to provide information to families. Nevertheless, better knowledge about the early and late predictive factors of long-term severe and moderate neurodevelopmental outcomes is badly needed.

This study is a prospective national observational population-based study involving all level III intensive care units in France.

This population-based cohort study will be performed including all moderate or severe cases of HIE, occurring between 34 and 42 completed weeks gestation in newborns admitted to a neonatal intensive care unit of the participating French regions. Children will be followed-up until the age of 3 years.

Participating centers will be invited to adhere to current HIE management guidelines and/or clinical investigations considered optimal to date, to ensure standardize clinical practice. The study will ensure high quality data collection.

About indications, timing and characteristics of treatments and investigations will be elaborated by the scientific committee during the preparation stage of the cohort study. This professional advice will have the double advantage of enabling us to record more homogeneous and high-quality data, and to standardize and improve clinical management and investigations among newborns with HIE.

Within this main study, an ancillary study will be performed by 21 centers to address the first secondary objective (predictive value of very early - first 6 hours of life - neurological examination and biological investigations, including specific new biomarkers such as Interleukin-6, Metalloproteinase-9, TIMP-1, Albumin modified by hypoxia, troponin I, acylcarnitins and amino acids).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at a gestational age of 34 weeks or more;
* Presenting early neurological distress with clinical signs of moderate to severe HIE at a standardized neurologic examination performed by a senior examiner:

  * Moderate HIE: lethargy, hyper-reflexia, miosis, bradycardia, seizures, hypotonia with weak suck and Moro reflex
  * Severe HIE: stupor, flaccidity, small to mid-position pupils that react poorly to light, reduced stretch reflexes, hypothermia or no Moro reflex
* With criteria for asphyxia:

  * pH of 7.0 or less or a base deficit of 16 mmol per liter or more in a sample of umbilical-cord blood or any blood sampled in the first hour after birth.
  * If, during this interval, the pH is between 7.01 and 7.15, base deficit is between 10 and 15.9 mmol per liter, or blood gas is not available, additional criteria will be required. These include:
  * an acute perinatal event (e.g., late or variable decelerations, cord prolapse, cord rupture, uterine rupture, maternal trauma, hemorrhage, or cardiorespiratory arrest)
  * or an abrupt change in fetal heart rate (FHR), defined as a persistent abnormal FHE after a period of normal tracing: bradycardia or prolonged deceleration, persistent variable decelerations, persistent late decelerations, and reduced heart variability
  * or either a 10-minute Apgar score of 5 or less or assisted ventilation initiated at birth and continued for at least 10 minutes.
* Written parental informed consent
* Covered by the French social security

Exclusion Criteria:

* Congenital malformations
* Chromosomal disorders
* Congenital neuromuscular disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be performed on all moderate or severe cases of hypoxic ischemic encephalopathyhie, occurring between 34 and 42 completed weeks gestation in newborns admitted to a neonatal intensive care unit of the participating French regions. Children will be followed-up until the age of 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is a combined criterion : death, neurodevelopmental disabilities in survivors | between birth and 3 years of age
  A combined criterion which includes:
  * Death between birth and 3 years of age
  * Neurodevelopmental disabilities in survivors, defined as :
    o Severe disabilities
  * Intellectual impairment with a mental score >2SD below the mean or <70 (ASQ)
  * Or Cerebral palsy with a Gross Motor Function level of 3-5 according to the GMFCS
  * Or bilateral blindness (vision <20/200 acuity)
  * Or deafness requiring amplification (>60dB)and/
  * Or a persistent disorder defined as recurrent seizures after discharge from neonatal intensive care requiring anti-convulsion therapy at the examination time point
    o Moderate disabilities
  * Intellectual impairment with a mental score >1SD below the mean or 70 to 84 (ASQ)
  * Cerebral palsy with a Gross Motor Function level of 1 or 2 according to the GMFCS
  * Or hearing impairment requiring no amplification

SECONDARY OUTCOMES:
First secondary objective : The relevance of specific new biomarkers : Protein levels (IL-6, MMP-9, TIMP-1, Albumine modified by hypoxia, troponine I), acylcarnitins and amino acids. | before H6 and at 3 days
  The biologist will evaluate the relevance of specific new biomarkers :
  * Protein levels (IL-6, MMP-9, TIMP-1, Albumine modified by hypoxia, troponine I) unites will be determined using an ELISA
  * the measurement of acylcarnitins and amino acids by tandem liquid phase chromatography coupled with mass spectroscopy.
  The analyses will be blinded and centralized to Reims University laboratory
Second secondary objective: the predictive value of clinical investigations during the first weeks of life and treatments. | first week, At 18 months and 3 years of age
  To analyze the predictive value of clinical investigations during the first weeks of life and treatments, including cooling:
  * for normal outcomes (absence of death, any disability, any epilepsy or any need for physiotherapy, orthophonist or psychologist or other measures of reeducation), moderate or severe neurodevelopmental disabilities, and death
  * At 18 months and 3 years of age
  * In this part, we will assess the ability of a normal developmental assessment at 18 months to predict survival free of disability or retardation at 3 years. This information will be useful in the future to define different strategies of follow up according to the assessment at 18 months of age.
Third secondary objective : Number and percentage of participants with cooling. | birth
  The third secondary objective is analyzed thanks to :
  * number of patients with method of cooling : Criticool, tecotherm, craft, other
  * duration of cooling in hours
  * number of severe or modere HIE according to the Sarnat classification
  * time to initiate cooling in minutes
Fourth secondary objective : Number and percentage of various obstetrical conditions leading to the worse outcomes | birth
  Number and percentage of :
  * Maternal pyrexia,
  * a persistent occipito-posterior position,
  * an acute intrapartum event (hemorrhage, maternal convulsions, rupture of uterus, snapped cord, and birth of baby before arrival at obstetric facility),
  * an instrumental vaginal delivery
  * an emergency caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DEBILLON, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (22):
- France (22):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - Chu Bordeaux, Bordeaux
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - CHU Clermond-Ferrand, Clermont-Ferrand
  - Chi Creteil, Créteil
  - Chu Dijon, Dijon
  - CHU FORT de France, Fort de France
  - Chu Grenoble, Grenoble
  - Chru Lille, Lille
  - Chu Limoges, Limoges
  - Chu Marseille, Marseille
  - CHU Montpellier, Montpellier
  - Chu La Miletrie, Poitiers
  - Chu Reims, Reims
  - Chu Rouen, Rouen
  - CHU St Denis, Saint-Denis de La Réunion
  - CHU St Pierre, Saint-Pierre
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- [Background] Volpe JJ. Neonatal encephalopathy: an inadequate term for hypoxic-ischemic encephalopathy. Ann Neurol. 2012 Aug;72(2):156-66. doi: 10.1002/ana.23647. PMID 22926849
- [Background] Use and abuse of the Apgar score. Committee on Fetus and Newborn, American Academy of Pediatrics, and Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Pediatrics. 1996 Jul;98(1):141-2. PMID 8668389
- [Background] Fenichel GM. Hypoxic-ischemic encephalopathy in the newborn. Arch Neurol. 1983 May;40(5):261-6. doi: 10.1001/archneur.1983.04050050029002. PMID 6405725
- [Background] Levene ML, Kornberg J, Williams TH. The incidence and severity of post-asphyxial encephalopathy in full-term infants. Early Hum Dev. 1985 May;11(1):21-6. doi: 10.1016/0378-3782(85)90115-x. PMID 4006822
- [Derived] Binet L, Debillon T, Beck J, Vilotitch A, Guellec I, Ego A, Chevallier M; LYTONEPAL research group. Effect of gestational age on cerebral lesions in neonatal encephalopathy. Arch Dis Child Fetal Neonatal Ed. 2024 Aug 16;109(5):562-568. doi: 10.1136/archdischild-2023-326131. PMID 38418209
- [Derived] Guellec I, Ancel PY, Beck J, Loron G, Chevallier M, Pierrat V, Kayem G, Vilotitch A, Baud O, Ego A, Debillon T. Glycemia and Neonatal Encephalopathy: Outcomes in the LyTONEPAL (Long-Term Outcome of Neonatal Hypoxic EncePhALopathy in the Era of Neuroprotective Treatment With Hypothermia) Cohort. J Pediatr. 2023 Jun;257:113350. doi: 10.1016/j.jpeds.2023.02.003. Epub 2023 Feb 23. PMID 36828343
- [Derived] Debillon T, Sentilhes L, Kayem G, Chevallier M, Zeitlin J, Baud O, Vilotitch A, Pierrat V, Guellec I, Ancel PY, Bednarek N, Ego A. Risk factors for unfavorable outcome at discharge of newborns with hypoxic-ischemic encephalopathy in the era of hypothermia. Pediatr Res. 2023 Jun;93(7):1975-1982. doi: 10.1038/s41390-022-02352-w. Epub 2022 Oct 22. PMID 36272997
- [Derived] Beck J, Debillon T, Guellec I, Vilotitch A, Loron G, Bednarek N, Ancel PY, Pierrat V, Ego A. Healthcare organizational factors associated with delayed therapeutic hypothermia in neonatal hypoxic-ischemic encephalopathy: the LyTONEPAL cohort. Eur J Pediatr. 2023 Jan;182(1):181-190. doi: 10.1007/s00431-022-04666-7. Epub 2022 Oct 21. PMID 36269426
- [Derived] Beck J, Bednarek N, Pierrat V, Vilotitch A, Loron G, Alison M, Guellec I, Hertz-Pannier L, de Launay C, Ego A, Vo-Van P, Ancel PY, Debillon T. Cerebral injuries in neonatal encephalopathy treated with hypothermia: French LyTONEPAL cohort. Pediatr Res. 2022 Sep;92(3):880-887. doi: 10.1038/s41390-021-01846-3. Epub 2021 Nov 20. PMID 34802036
- [Derived] Debillon T, Bednarek N, Ego A; LyTONEPAL Writing Group. LyTONEPAL: long term outcome of neonatal hypoxic encephalopathy in the era of neuroprotective treatment with hypothermia: a French population-based cohort. BMC Pediatr. 2018 Aug 1;18(1):255. doi: 10.1186/s12887-018-1232-6. PMID 30068301